CLINICAL TRIAL: NCT00785083
Title: A Double-blind, Randomized, Placebo-controlled, Parallel, Time-lagged, Ascending, Multi-centre, Multiple-dose Study to Measure the Magnitude and Time Course of the Effect of FTY720 on FEV1 and Other Pulmonary Function Tests (FVC, FEF25-75%, and FEV1/FVC) in Patients With Moderate Asthma
Brief Title: A Study of the Effect of FTY720 on Pulmonary Function in Patients With Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFTY720D2102
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Asthma, adrenergic beta agonists, multiple sclerosis, pulmonary function tests, forced expiratory volume
MeSH Terms: conditions — Asthma; Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: FTY720
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FTY720
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will evaluate the effect of FTY720 on the lung function of patients with moderate asthma

ELIGIBILITY:
Inclusion Criteria:

* Forced Expiratory Volume in 1 second of at least 60%
* History of asthma for at least 6 months
* Current use of short-acting beta agonists, inhaled long-acting beta agonists and inhaled corticosteroids (up to a specified dose)

Exclusion Criteria:

* History of lung disease other than asthma
* Smokers
* Use of inhaled corticosteroid above specified dose
* Use of oral beta agonists or corticosteroids or other asthma medications
* Hypersensitivity to the drug
* Respiratory tract infections within 1 month of the study

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pulmonary function tests (particularly Forced Expiratory Volume at 1 sec (FEV1) at Day 10 | 10 days
Safety of FTY720 | 10 days

SECONDARY OUTCOMES:
Use of short acting beta agonists during treatment compared to pre-treatment | 10 days
Pharmacokinetics of FTY720 and FTY720-P | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis Investigator Site
Locations (1):
- Novartis Investigator Site, Manchester, United Kingdom

REFERENCES:
- [Result] Boulton C, David OJ, Meiser K, Schmouder R. Tolerability and Pulmonary Pharmacodynamic Effects During Treatment Initiation of Once-Daily Oral Fingolimod in Subjects With Moderate Asthma. Clin Pharmacol Drug Dev. 2013 Jan;2(1):2-10. doi: 10.1002/cpdd.4. Epub 2013 Mar 4. PMID 27121555
- [Derived] Izquierdo G, O'Connor P, Montalban X, von Rosenstiel P, Cremer M, de Vera A, Sfikas N, Francis G, Radue EW, Kappos L. Five-year results from a phase 2 study of oral fingolimod in relapsing multiple sclerosis. Mult Scler. 2014 Jun;20(7):877-81. doi: 10.1177/1352458513513059. Epub 2013 Nov 30. PMID 24293455